CLINICAL TRIAL: NCT00282386
Title: A Multicenter, Randomized, Parallel-Group, Placebo-Controlled, Double-Blind Study With In-House Blinding to Determine the Effect of 156 Weeks of Treatment With MK0966 on the Recurrence of Neoplastic Polyps of the Large Bowel in Patients With a History of Colorectal Adenomas
Brief Title: A Study to Evaluate the Effect of MK0966 (Rofecoxib) on the Recurrence of Colorectal Adenomas (0966-122)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 0966-122; 2006_005
Record Dates: First submitted 2006-01-24; First posted 2006-01-26 (Estimated); Last update posted 2017-05-09 (Actual); Status verified 2017-05

CONDITIONS: Colorectal Adenoma
MeSH Terms: interventions — rofecoxib; Duration of Therapy

STUDY DESIGN:
Who Masked: Participant, Investigator

INTERVENTIONS:
Drug: MK0966; Rofecoxib / Duration of Treatment: 156 weeks
Drug: Placebo/ Duration of Treatment: 156 weeks

SUMMARY:
This study was to compare the effect of 156 weeks of treatment with MK-0966 (Rofecoxib) versus placebo on the recurrence of colorectal adenomas (growths that occur on the inside (the lining) of the large intestine, also known as the colon) in patients with a history of colorectal adenomas.

ELIGIBILITY:
Inclusion Criteria:

* Eligible patients must have undergone a complete colonoscopy within 12 weeks of study entry with removal of all polyps; at least one polyp must have been confirmed a large bowel pre-cancerous polyp (adenoma) by the study pathologist.

Exclusion Criteria:

* History with a specific hereditary large bowel polyp syndrome
* History of a large bowel adenoma before age 35
* Small or large bowel resection or history of inflammatory bowel disease
* History of cancer within the five years before enrollment
* Expected need for chronic NSAID therapy
* Positive test result for stool occult blood
* Uncontrolled hypertension, stroke or temporary mini stroke (TIA) within the past 2 years, angina or congestive heart failure with symptoms that occur at rest or with minimal activity
* History of myocardial infarction (heart attack), coronary angioplasty, or coronary artery bypass grafting within the past 1 year
* Pregnancy

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2586 (Actual)
Dates: Start 1999-12-23 (Actual); Primary Completion 2004-09-01 (Actual); Study Completion 2004-09-01 (Actual)

PRIMARY OUTCOMES:
Cumulative colorectal adenoma recurrence during treatment in patients with an increased risk to develop colorectal cancer. | 156 Weeks

SECONDARY OUTCOMES:
Cumulative colorectal adenoma recurrence during treatment in patients with a history of colorectal adenoma | 156 Weeks
Cumulative colorectal adenoma recurrence during treatment in all patients | 52 Weeks
To evaluate safety & tolerability of rofecoxib

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

REFERENCES:
- [Background] Bresalier RS, Sandler RS, Quan H, Bolognese JA, Oxenius B, Horgan K, Lines C, Riddell R, Morton D, Lanas A, Konstam MA, Baron JA; Adenomatous Polyp Prevention on Vioxx (APPROVe) Trial Investigators. Cardiovascular events associated with rofecoxib in a colorectal adenoma chemoprevention trial. N Engl J Med. 2005 Mar 17;352(11):1092-102. doi: 10.1056/NEJMoa050493. Epub 2005 Feb 15. PMID 15713943
- [Background] Baron JA, Sandler RS, Bresalier RS, Quan H, Riddell R, Lanas A, Bolognese JA, Oxenius B, Horgan K, Loftus S, Morton DG; APPROVe Trial Investigators. A randomized trial of rofecoxib for the chemoprevention of colorectal adenomas. Gastroenterology. 2006 Dec;131(6):1674-82. doi: 10.1053/j.gastro.2006.08.079. Epub 2006 Sep 1. PMID 17087947
- [Background] Lanas A, Baron JA, Sandler RS, Horgan K, Bolognese J, Oxenius B, Quan H, Watson D, Cook TJ, Schoen R, Burke C, Loftus S, Niv Y, Ridell R, Morton D, Bresalier R. Peptic ulcer and bleeding events associated with rofecoxib in a 3-year colorectal adenoma chemoprevention trial. Gastroenterology. 2007 Feb;132(2):490-7. doi: 10.1053/j.gastro.2006.11.012. Epub 2006 Nov 10. PMID 17258718
- [Derived] Baron JA, Sandler RS, Bresalier RS, Lanas A, Morton DG, Riddell R, Iverson ER, Demets DL. Cardiovascular events associated with rofecoxib: final analysis of the APPROVe trial. Lancet. 2008 Nov 15;372(9651):1756-64. doi: 10.1016/S0140-6736(08)61490-7. Epub 2008 Oct 14. PMID 18922570
- Available data/document: CSR Synopsis — http://www.merck.com/clinical-trials/policies-perspectives.html